CLINICAL TRIAL: NCT01396486
Title: A Randomized Controlled Trial of Inositol and Omega-3 Fatty Acids in Pediatric Mania
Brief Title: Inositol and Omega-3 Fatty Acids in Pediatric Mania
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Janet Wozniak, MD, Assistant Professor of Psychiatry at Harvard Medical School and at Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-P-001937
Record Dates: First submitted 2011-07-15; First posted 2011-07-18 (Estimated); Results first posted 2020-04-21 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Pediatric Bipolar Spectrum Disorders
Keywords: Omega-3 Fatty Acids; Fish Oil; Inositol; Natural supplements; Bipolar Spectrum Disorders; Mania; Depression; Children
MeSH Terms: conditions — Mania; Depression | interventions — Docosahexaenoic Acids; Inositol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Omega-3/Placebo (Active Comparator): Combination Omega-3 and Placebo treatment.
  Interventions: Drug: Omega-3
- Placebo/Inositol (Active Comparator): Combination Placebo and Inositol treatment.
  Interventions: Drug: Inositol
- Omega-3/Inositol (Active Comparator): Combination Omega-3 and Inositol treatment.
  Interventions: Drug: Omega-3; Drug: Inositol

INTERVENTIONS:
Drug: Omega-3 — Children with bipolar spectrum disorders ages 6-12 will receive treatment with omega-3 fatty acids. Study subjects may be randomized to receive 3000mg (6 500mg capsules) of omega-3 fatty acids for the duration of the study. Omega-3 fatty acid capsules are in the form of Nordic Naturals brand, ProOmega Junior, which contains 325mg EPA and 225mg DHA per two capsules.
  Other Names: ProOmega Junior
  Arms: Omega-3/Inositol; Omega-3/Placebo
Drug: Inositol — Children with bipolar spectrum disorders ages 6-12 will receive treatment with inositol, omega-3 fatty acids, or both weekly for 12 weeks. Subjects weighing 25kg or more may be randomized to receive 2000mg (4 500mg capsules) of inositol (80mg/kg for a 25kg child). Children weighing less than 25kg will be dosed at 80mg/kg rounded down to the nearest thousand mg dose. Dosage will remain constant throughout the study.
  Arms: Omega-3/Inositol; Placebo/Inositol

SUMMARY:
The purpose of this study is to a) evaluate the efficacy of omega-3 fatty acids versus inositol in the treatment of pediatric bipolar disorder, b) evaluate the efficacy of omega-3 fatty acid plus inositol in the treatment of pediatric bipolar disorder, and c) assess the side effect profile of omega-3 fatty acids plus inositol. This study will be a 12-week trial with children ages 5-12 years old with bipolar spectrum disorders.

DETAILED DESCRIPTION:
The investigators propose to conduct a randomized, double blind, controlled trial that will evaluate effectiveness and tolerability of omega-3 fatty acids and inositol used alone and in combination. The investigators plan to decrease the variability in the population under study by limiting the age range to 5-12 years and excluding cases with significant, untreated, comorbidity. The cognitive effects/side effects with a neuropsychological battery pre and post treatment will be measured. Subjects with a history of failing treatment with two or more conventional treatments will be excluded.

This will be a 12-week, double-blind, randomized clinical trial study to compare efficacy and tolerability of the natural treatments omega-3 fatty acids and inositol used in combination in the treatment of bipolar spectrum disorders in children and adolescents (ages 5-12). Subjects will be randomized in double blind fashion to one of three arms: omega-3 fatty acids, inositol or the combined treatment. Further, the proposed study will include measures of cognition prior to starting study medication and at endpoint. The investigators will minimize the variability of the population under study by limiting the age range to 5-12 years, minimizing untreated or clinically significant comorbidity and excluding subjects who have already failed treatment with 2 or more anti-manic agents. Subjects will include youth ages 5-12 years with a bipolar spectrum disorder (type I, II, or NOS), mixed, manic, or hypomanic state, according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (American Psychiatric Association, 2000) (DSM-IV), randomized to 3 treatment arms: 1) treatment with omega-3 fatty acids (N=20); 2) treatment with inositol (N=20); 3) treatment with the combination of inositol and omega-3 fatty acids (N=20).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 5-12 years of age.
2. Subjects must have a DSM-IV diagnosis of a bipolar spectrum disorder (type I, II, or Not Otherwise Specified (NOS)), and currently displaying mixed, manic, or hypomanic symptoms (without psychotic features) according to the DSM-IV based on clinical assessment and confirmed with structured diagnostic interview (Schedule of Affective Disorders and Schizophrenia for School-Age Children - Epidemiological Version (K-SADS-E)) (Orvaschel, 1994).
3. Subjects and their legal representative must have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
4. Subjects and their legal representative must be considered reliable.
5. Each subject and his/her authorized legal representative must understand the nature of the study. The subject's authorized legal representative must sign an informed consent document and the subject must sign an informed assent document.
6. Subjects must have an initial score on the YMRS total score of at least 20.
7. Subject must be able to swallow pills.
8. Subjects with ADHD and ODD will be allowed to participate in the study provided that the impairment associated with these disorders is of mild or moderate severity (not severe) and milder in severity relative to the impairment of the bipolar disorder, according to clinician evaluation. Subjects with comorbid anxiety disorders will be allowed to participate provided that the impairment associated with the anxiety is of minimal severity, according to clinician evaluation. Subjects with comorbid CD will be excluded.

Exclusion Criteria:

1. Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild.
2. Serious or unstable illness including hepatic, renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
3. History of bleeding diathesis, including those with von Willebrand disease.
4. Uncorrected hypothyroidism or hyperthyroidism.
5. History of sensitivity to omega-3 fatty acids or inositol. A non-responder or history of intolerance to omega-3 fatty acid or inositol, after 2 months of treatment at adequate doses as determined by the clinician.
6. Severe allergies or multiple adverse drug reactions.
7. Failed 2 or more previous trials with anti-manic treatments including lithium, anticonvulsants and atypical antipsychotic medication.
8. Current or past history of seizures.
9. DSM-IV substance use, abuse or dependence (unlikely in ages 5-12).
10. Judged clinically to be at serious suicidal risk.
11. Current diagnosis of schizophrenia.
12. Current diagnosis of conduct disorder
13. Pregnancy (unlikely in ages 5-12).
14. YMRS Item #8 (Content) score of 8 ("delusions; hallucinations").
15. YMRS total score above 40.
16. Girls who have begun menstruating.
17. C-SSRS score ≥ 4.
18. IQ < 70.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2012-02-03 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Wozniak, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wozniak J, Faraone SV, Chan J, Tarko L, Hernandez M, Davis J, Woodworth KY, Biederman J. A randomized clinical trial of high eicosapentaenoic acid omega-3 fatty acids and inositol as monotherapy and in combination in the treatment of pediatric bipolar spectrum disorders: a pilot study. J Clin Psychiatry. 2015 Nov;76(11):1548-55. doi: 10.4088/JCP.14m09267. PMID 26646031

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While 69 subjects enrolled in the study, only 61 were randomized. Of the 8 subjects who enrolled but were not randomized, 3 were found ineligible, 3 withdrew, and 2 were lost to follow-up.
Period: Overall Study
Arm/Group | Omega-3/Placebo | Placebo/Inositol | Omega-3/Inositol
Started | 20 | 19 | 22
Exposed | 19 | 16 | 17
Completed | 10 | 7 | 10
Not Completed | 10 | 12 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega-3/Placebo | Placebo/Inositol | Omega-3/Inositol | Total
Number analyzed (Participants) | 19 | 16 | 17 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.8 (1.6) | 8.8 (2.3) | 8.4 (2.5) | 8.3 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 8 | 20
  Male | 11 | 12 | 9 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 0 | 6
  Not Hispanic or Latino | 14 | 14 | 17 | 45
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 16 | 14 | 16 | 46
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 19 | 16 | 17 | 52
YMRS [Mean (Standard Deviation); unit: units on a scale] — The Young Mania Rating Scale (YMRS) consists of 7 items rated on a scale from 0 (symptoms not present) to 4 (symptoms extremely severe) and 4 items rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe).The YMRS score ranges from 0-60. Questions are asked about the last week. A higher score signifies more severe manic symptoms.
  units on a scale | 26.1 (7.2) | 25.8 (6.5) | 24.2 (5.8) | 25.4 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Mania Symptoms by Change in Young Mania Rating Scale (YMRS)
Description: The Young Mania Rating Scale (YMRS) consists of 7 items rated on a scale from 0 (symptoms not present) to 4 (symptoms extremely severe) and 4 items rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe).The YMRS score ranges from 0-60. Questions are asked about the last week. A higher score signifies more severe manic symptoms.
Time Frame: Baseline to endpoint (12 weeks or last observation carried forward if dropped prior to week 12)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omega-3/Placebo | Placebo/Inositol | Omega-3/Inositol
Number analyzed (Participants) | 19 | 16 | 17
units on a scale | -4.8 (7.9) | -6.4 (6.4) | -10.2 (9.0)

2. Primary Outcome: Improvement in Depression Symptoms by Children's Depression Rating Scale (CDRS)
Description: The Children's Depression Rating Scale (CDRS) is a clinician-rated instrument with 17 items scored on a 1 to 5 or 1 to 7 scale. A rating of 1 indicates normal, thus the minimum score is 17. The maximum score is 113. Scores of 20-30 suggest borderline depression. Scores of 40-60 indicate moderate depression.
Time Frame: Baseline to endpoint (12 weeks or last observation carried forward if dropped prior to week 12)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omega-3/Placebo | Placebo/Inositol | Omega-3/Inositol
Number analyzed (Participants) | 19 | 16 | 17
units on a scale | -4.9 (10.6) | -5.6 (10.1) | -10.8 (7.4)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Consistent with good clinical practice, safety will be monitored by each subject's study clinician at each study visit. Subjects will be monitored by the study clinician for adverse events at each visit and adverse events will be recorded on an Adverse Events Form.
Arm/Group | Omega-3/Placebo | Placebo/Inositol | Omega-3/Inositol
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/19 | 0/22
Other Adverse Events (participants affected / at risk) | 13/20 | 12/19 | 10/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3/Placebo (N=20) | Placebo/Inositol (N=19) | Omega-3/Inositol (N=22)
Agitated/Irritable (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) — Required ER visit.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omega-3/Placebo (N=20) | Placebo/Inositol (N=19) | Omega-3/Inositol (N=22)
Nausea/Vomit/Diarrhea (Gastrointestinal disorders) | 4 | 1 | 3
Cold/Infection/Allergy (Infections and infestations) | 3 | 1 | 1
Agitated/Irritable (Psychiatric disorders) | 1 | 2 | 0
Headache (General disorders) | 0 | 1 | 1
Insomnia (Nervous system disorders) | 0 | 1 | 1
Sedation (Nervous system disorders) | 0 | 1 | 0
Tics (Psychiatric disorders) | 0 | 0 | 1
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Increased Appetite (General disorders) | 0 | 2 | 1
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatological (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Thirsty (General disorders) | 0 | 0 | 1
Dizzy/Lightheaded (General disorders) | 0 | 0 | 1
Bet Wetting (General disorders) | 1 | 0 | 0
Earache (Ear and labyrinth disorders) | 0 | 0 | 1
Irregular Behavior (General disorders) | 1 | 0 | 0
Weight Gain (General disorders) | 0 | 1 | 0
Neurological (Nervous system disorders) | 0 | 0 | 1
Autonomic (Nervous system disorders) | 0 | 0 | 1
Strep Throat (Infections and infestations) | 1 | 0 | 0
Psychotic Episode (Psychiatric disorders) | 0 | 1 | 0
Sleep Walking (Nervous system disorders) | 0 | 1 | 0
Scrape (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chewing Inside of Cheek (General disorders) | 0 | 1 | 0
Agitated with Homicidal Statements (Psychiatric disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/86/NCT01396486/Prot_SAP_000.pdf